CLINICAL TRIAL: NCT05680519
Title: Preventing Non-communicable Diseases by Screening and Educating Emergency Department Attendees on Health-risk Behaviours: A Pilot Randomized Controlled Trial
Brief Title: Screening and Educating Emergency Department Attendees on Health-risk Behaviours
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Ho Cheung William, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.565
Record Dates: First submitted 2022-12-02; First posted 2023-01-11 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Health-risk Behaviours; Non Communicable Diseases
Keywords: Health-risk Behaviours; Non Communicable Diseases; Emergency Department
MeSH Terms: conditions — Noncommunicable Diseases; Emergencies | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants will also be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications. The participants will receive a brief telephone intervention using the Ask, Warn, Advise, Refer and Do-it-again (AWARD) model. For the advice step, the research assistant will ask about the priority the participants place on engagement in desirable health-related lifestyle practices identified in the completed behavioural risk factor survey. The participants will also be asked to choose the goal that they consider easiest to achieve, such as quitting or reducing smoking, consuming more vegetables or less fatty foods or sugary drinks, performing more exercise or reducing alcohol consumption. The participants will be encouraged to quit health-risk behaviours (or adopt a healthy lifestyle) sequentially, but they will also be able to choose to quit them simultaneously if they are confident in doing so.
  Interventions: Other: theory of planned behaviour, foot-in-the-door technique, and self-determination theory intervention
- Control group (Placebo Comparator): The participants will also be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications. The control group participants will receive a brief telephone intervention based on the AWARD model and delivered by the trained research assistant, similar to that delivered to the intervention group. However, the research assistant will simply advise the participants to modify their health-risk behaviours and/or adopt a healthy lifestyle practice. In addition, the research assistant will send regular SMS messages to the participants at a similar frequency to the intervention group, but these messages will contain only general health advice. The participants will also receive follow-up for outcome assessments with the same schedule as those in the intervention group.
  Interventions: Other: Control group

INTERVENTIONS:
Other: theory of planned behaviour, foot-in-the-door technique, and self-determination theory intervention — The participants will also be asked to choose the goal that they consider easiest to achieve and encouraged to quit health-risk behaviours. The research assistant will assist in achieving the participant's health-related goals by sending WhatsApp/WeChat messages or via telephone calls once per week for the first 6 months.
  Arms: Intervention group
Other: Control group — The participants will be simply advised to modify their health-risk behaviours and/or adopt a healthy lifestyle practice. In addition, the research assistant will send regular SMS messages to the participants at a similar frequency to the intervention group, but these messages will contain only general health advice.
  Arms: Control group

SUMMARY:
Aim:

To determine the feasibility and potential efficacy of a proactive approach using a brief self-determination theory-based intervention to help people attending the ED modify their health-risk behaviours and lead healthier lives.

Objectives

1. To assess the recruitment, participation and retention rates of targeted participants in an emergency department
2. To ascertain the feasibility of screening, recruiting and educating people to change health-risk behaviours in the emergency department

DETAILED DESCRIPTION:
Setting:

The setting is the ED of the United Christian Hospital (UCH), one of the major acute care hospitals in Kowloon East cluster in Hong Kong.

Intervention:

At the ED The potential participants will first be invited by our research assistant to complete a baseline behavioural risk factor survey. Those whose survey responses indicate that they are eligible participants will be explained the purpose and nature of the study and will be asked to sign an informed consent form. They will then be informed that they will receive a telephone call from a research assistant within 3 days to evaluate their assessment outcomes and provide them with appropriate interventions. The participants will also be given a Practical Resource Hub for Healthy Life leaflet containing information on various applications, including (i) 'Move Your Body', (ii) 'Eat Healthy', (iii) 'Live Alcohol Free', and (iv) 'Stay Away from Tobacco', which were developed by the Hong Kong Department of Health.

1. Intervention group Brief intervention via telephone (within 3 days after visiting the ED) The participants will receive a brief intervention using the Ask, Warn, Advise, Refer and Do-it-again (AWARD) model, which was originally developed for primary-care tobacco-cessation interventions. The brief intervention includes the following steps: (1) ask about and assess health-risk behaviours; (2) warn about the high morbidity and mortality risks associated with health-risk behaviours; (3) advise to adopt healthy lifestyle practices to benefit the health of the participant; (4) refer to hotline services on request, such as smoking cessation and alcohol treatment services; and (5) do it again. For the warning message, the research assistant will provide the following standardised message: 'The WHO has identified four major behavioural risk factors, namely, tobacco use, harmful alcohol use, an unhealthy diet and physical inactivity, that contribute substantially to NCDs, which result in high rates of morbidity and mortality.' For the advice step, the research assistant will ask about the priority the participants place on engagement in desirable health-related lifestyle practices identified in the completed behavioural risk factor survey. The participants will also be asked to choose the goal that they consider easiest to achieve, such as quitting or reducing smoking, consuming more vegetables or less fatty foods or sugary drinks, performing more exercise or reducing alcohol consumption. The participants will be encouraged to quit health-risk behaviours (or adopt a healthy lifestyle) sequentially, but they will also be able to choose to quit them simultaneously if they are confident in doing so. Each participant will then receive a brief (approximately 5 minutes), individual intervention with health advice about the selected health-related lifestyle practice. The whole intervention will last approximately 10 minutes, but slightly longer if necessary. Such a brief intervention will be cost-effective and more feasible for routine use in clinical practice by healthcare professionals after minimal training. Previous clinical trials of smoking cessation have provided strong evidence regarding the effectiveness of brief interventions using the AWARD model.

   At the end of the telephone call, the participants will be informed that throughout the study period, the research assistant will assist in achieving the participant's health-related goals by sending WhatsApp/WeChat messages or via telephone calls.

   Follow-up booster intervention (up to 6 months) For the first 6 months of the study period, the research assistant will deliver WhatsApp/WeChat messages about once per week. If a participant does not own a smartphone or is unable to receive WhatsApp/WeChat messages (uncommon in Hong Kong), the research assistant will make a telephone call, instead of sending a message, as a reminder for the participants to adhere to their desirable health-related lifestyle practice. Instant messaging via mobile applications has found to be effective in enhancing treatment compliance.

   Follow-up assessment of behavioural changes at 3, 6, and 12 months The participants will be assessed to determine their success in changing their targeted health-related lifestyle practice via a phone call at 3, 6, and 12 months.
2. Control group The control group participants will receive a brief telephone intervention based on the AWARD model and delivered by the trained research assistant, similar to that delivered to the intervention group. However, the research assistant will simply advise the participants to modify their health-risk behaviours and/or adopt a healthy lifestyle practice. In addition, the research assistant will send regular SMS messages to the participants at a similar frequency to the intervention group, but these messages will contain only general health advice. The participants will also receive follow-up for outcome assessments with the same schedule as those in the intervention group.

(i) Study design A pilot RCT with a two-group pre-test and repeated post-test between- subjects design will be conducted.

Subject recruitment The investigators will obtain ethical approval from the institutional review board of the Kowloon East cluster. Potential participants will be assessed for eligibility, and the purpose, design, procedures, and potential benefits and risks of the study will be explained to them. Informed written consent will then be sought. All subjects will be assured that their participation will be voluntary, with no prejudice attached to refusal, and that the information they provide will be kept confidential. The researcher is responsible for its safekeeping and the only one who would have access to the raw data or study record during or after the study. After the period of storage, all raw data and records will be destroyed.

The proposed study will adhere to the Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Subjects.

Randomization and allocation concealment To avoid the potential risk of treatment contamination within the ED, randomisation will not be performed there. Instead, the research assistant will input the baseline data collected at the ED directly into the web-based trial entry form linked to a computerised database, and randomisation will then be performed at the Principal Investigator's (PI's) institution by an independent statistician who will have no other involvement in the study. Stratified block randomisation with 1:1 allocation will be conducted using varying block sizes of 2-4 to achieve an appropriate balance of participant numbers between the two groups and to optimise allocation concealment.

(ii) Data processing and analysis

Instruments:

A behavioural risk-factor survey will be used to collect the eligible participants' demographic and clinical data and information about their health-risk behaviours at baseline and at 3, 6, and 12 months. This questionnaire is adapted from a questionnaire used by the Hong Kong Department of Health and was used to investigate multiple health-risk behaviours among Chinese adults in Hong Kong in 2021.

The EuroQoL 5-Dimension 5-level (EQ-5D-5L) will be used to measure subjects' health-related quality of life at baseline, 6 months, and 12 months. The psychometric properties of the Chinese version of the EQ-5D-5L have been tested, and the findings indicate that this tool is a valid, reliable, and sensitive measure of health-related quality of life. A Chinese-specific EQ-5D-5L value set will enable the estimation of health utility scores applicable to the Chinese population and quality-adjusted life-years (QALY) for cost-effectiveness analysis (CEA).

All the baseline data will be collected by a research assistant during the daytime. In addition, details of the study, consent form and information sheet, and the questionnaire will be installed on tablet computers and hung on the wall in a prominent place of the ED. In the absence of the research assistant, anyone who wants to participate in the health risk screening can do it themselves through the tablet computers. The tablet is user friendly. Furthermore, such systems have built-in functions to protect against errors and allow the collected data to be easily processed for progress monitoring and analysis. A research assistant will then contact subjects by phone and provide them with health-related lifestyle advice and follow-up.

Sample size:

The investigators identified no similar randomised controlled trials (RCTs) in PubMed, Cochrane Library or clinical trial registries (ClinicalTrials.gov and ISRCTN). The investigators therefore used G*Power to estimate the sample size based on the results of a previous study on testing the efficacy of a self-determination theory-based smoking cessation intervention for smokers at emergency departments. The results showed that the intervention was effective in helping people quit smoking at 12-month follow-up (RR = 1.46 [95%CI = 1.06-2.19]). To detect a significant between-group difference with a power of 80% at a significance level of 5% (two-tailed) in the proportion of participants changing their health-risk behaviours, 501 participants will be needed per group. To account for a potential attrition rate of 30% at the 12-month follow-up, a total of 1,431 participants will be required for a full scale RCT.

For the sample size of the pilot study, the investigators use the recommendation of at least 10% of the sample required for a full study recommended by Hertzog. Accordingly, 150 participants will be targeted for this pilot study. Based on daily attendance information from UCH's Chief of Service in-charge and the nurse consultant working at A&E, the investigators are confident that the required number of participants can be recruited within 6 months.

Data Analysis:

The baseline characteristics of the two groups will first be compared using the chi-square test for categorical variables and analysis of variance for continuous variables. Intention-to-treat analysis will be used by imputing all non-responses at follow-up by baseline values (i.e. assuming failure or no change after the intervention), to yield more conservative effect size estimates. For the qualitative interview, the data analysis process will begin immediately after each individual interview, in accordance with the thematic analysis framework introduced by Braun and Clarke, using NVivo version 12 (2018; QSR International Pty Ltd, Melbourne, Australia). The codes, categories and themes generated by this process will be compared.

SPSS for Windows (SPSS version 26.0; IBM Corp., Armonk, NY, USA) will be used for the quantitative data analysis. Descriptive statistics will be used to calculate the mean, standard deviation, and frequency of the demographic and health-risk behaviour data. The analysis including the main effect, i.e., behavioural changes at 12 months in the intervention group versus those in the control group, will be performed using a chi-square test or Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≥18 years,
* (2) triage as semi-urgent (level 4) or non-urgent (level 5), and
* (3) the presence of at least one health risk behaviour (tobacco use, harmful use of alcohol, unhealthy diet and physical inactivity)

Exclusion Criteria:

* (1) poor cognitive state or mental illness and
* (2) participation in another related study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study | at baseline
  Assess the feasibility of the study through the recruitment/participation rate
Feasibility of the study | 3 months
  Assess the feasibility of the study through the participation/retention rate
Feasibility of the study | 6 months
  Assess the feasibility of the study through the participation/retention rate
Feasibility of the study | 12 months
  Assess the feasibility of the study through the participation/retention rate

SECONDARY OUTCOMES:
Change of smoking consumption | 3 months
  The participants' change of smoking consumption between baseline and 3 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of tobacco product. The more frequencies and the more kinds of tobacco product used to indicate the higher smoking consumption.
Change of smoking consumption | 6 months
  The participants' change of smoking consumption between baseline and 6 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of tobacco product. The more frequencies and the more kinds of tobacco product used to indicate the higher smoking consumption.
Change of smoking consumption | 12 months
  The participants' change of smoking consumption between baseline and 12 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of tobacco product. The more frequencies and the more kinds of tobacco product used to indicate the higher smoking consumption.
Change of alcohol consumption | 3 months
  The participants' change of alcohol consumption between baseline and 3 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of alcohol product. The more frequencies and the more kinds of alcohol product used to indicate the higher alcohol consumption.
Change of alcohol consumption | 6 months
  The participants' change of alcohol consumption between baseline and 6 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of alcohol product. The more frequencies and the more kinds of alcohol product used to indicate the higher alcohol consumption.
Change of alcohol consumption | 12 months
  The participants' change of alcohol consumption between baseline and 12 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of alcohol product. The more frequencies and the more kinds of alcohol product used to indicate the higher alcohol consumption.
Change of physical inactivity | 3 months
  The participants' change of physical activity between baseline and 3 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of physical activity. The more frequencies and the more kinds of physical activity used to indicate the greater amount of physical activity.
Change of physical inactivity | 6 months
  The participants' change of physical activity between baseline and 6 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of physical activity. The more frequencies and the more kinds of physical activity used to indicate the greater amount of physical activity.
Change of physical inactivity | 12 months
  The participants' change of physical activity between baseline and 12 months follow-up using a Structured-Questionnaire gathering the frequency and kinds of physical activity. The more frequencies and the more kinds of physical activity used to indicate the greater amount of physical activity.
Change of unhealthy diet | 3 months
  The participants' change of unhealthy diet between baseline and 3 months follow-up using a Structured-Questionnaire gathering the frequency and amount of vegetable and fruit. The low frequencies and the low amount of vegetable and fruit used to indicate more unhealthy diet.
Change of unhealthy diet | 6 months
  The participants' change of unhealthy diet between baseline and 6 months follow-up using a Structured-Questionnaire gathering the frequency and amount of vegetable and fruit. The low frequencies and the low amount of vegetable and fruit used to indicate more unhealthy diet.
Change of unhealthy diet | 12 months
  The participants' changes of unhealthy diet between baseline and 12 months follow-up using a Structured-Questionnaire gathering the frequency and amount of vegetable and fruit. The low frequencies and the low amount of vegetable and fruit used to indicate more unhealthy diet.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project has been completed and the results of the project has been published
Access Criteria: Request could be sent to Principal Investigator (williamli@cuhk.edu.hk)